CLINICAL TRIAL: NCT03474094
Title: A European, Multicenter, Randomized, Open-label, Phase II Trial Aiming to Assess the Clinical and Biological Activity of an Anti-PD-L1 (Atezolizumab) in Operable Localised Soft Tissue Sarcomas Patients to be Treated With Radiotherapy
Brief Title: Clinical and Biological Activity of an Anti-PD-L1 (Atezolizumab) in Operable Localised Soft Tissue Sarcomas Patients to be Treated With Radiotherapy
Acronym: RT-Immune
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RT-Immune (ET16-132)
Record Dates: First submitted 2018-03-06; First posted 2018-03-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Sarcoma,Soft Tissue
Keywords: Clinical Trial; randomized; phase II; atezolizumab; PD-L1
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pre-operative radiotherapy and atezolizumab (Experimental): Pre-operative radiotherapy followed by 2 cycles of atezolizumab then surgery
  Interventions: Combination Product: Pre-operative radiotherapy followed by 2 cycles of atezolizumab then surgery
- pre-operative atezolizumab and post-operative radiotherapy (Experimental): 2 cycles of atezolizumab followed by surgery then post-operative radiotherapy
  Interventions: Combination Product: 2 cycles of atezolizumab followed by surgery then post-operative radiotherapy
- pre-operative radiotherapy and post-operative atezolizumab (Active Comparator): Pre-operative radiotherapy then surgery followed by 2 cycles of atezolizumab
  Interventions: Combination Product: Pre-operative radiotherapy followed by surgery then 2 cycles of atezolizumab.

INTERVENTIONS:
Combination Product: Pre-operative radiotherapy followed by 2 cycles of atezolizumab then surgery — W1,W2, W3, W4 & W5: RADIOTHERAPY. A 3-dimensional conformal RT (3D-CRT) with photons ≥ 6MV will be realized based on the acquisition of a CT-scan performed in treatment position. Intensity modulated RT (IMRT), volumetric modulated arc therapy (VMAT) and tomotherapy are authorized.
  W6 and W9: ATEZOLIZUMAB IV INJECTION. 2 injections of 1200 mg of atezolizumab with a 3-week interval
  W11: SURGERY. Surgery should be performed as per Institutional practice by a surgeon with appropriate training in the treatment of sarcoma. The primary aim of surgery is to completely excise the tumor with a margin of normal tissue commonly accepted as 1 cm soft tissue, or equivalent
  Arms: pre-operative radiotherapy and atezolizumab
Combination Product: 2 cycles of atezolizumab followed by surgery then post-operative radiotherapy — W1 and W4: ATEZOLIZUMAB IV INJECTION. 2 injections of 1200 mg of atezolizumab with a 3-week interval
  W6: SURGERY Surgery should be performed as per Institutional practice by a surgeon with appropriate training in the treatment of sarcoma. The primary aim of surgery is to completely excise the tumor with a margin of normal tissue commonly accepted as 1 cm soft tissue, or equivalent
  W7, W8, W9, W10 & W11: RADIOTHERAPY A 3-dimensional conformal RT (3D-CRT) with photons ≥ 6MV will be realized based on the acquisition of a CT-scan performed in treatment position. Intensity modulated RT (IMRT), volumetric modulated arc therapy (VMAT) and tomotherapy are authorized.
  Arms: pre-operative atezolizumab and post-operative radiotherapy
Combination Product: Pre-operative radiotherapy followed by surgery then 2 cycles of atezolizumab. — W1,W2, W3, W4 & W5: RADIOTHERAPY A 3-dimensional conformal RT (3D-CRT) with photons ≥ 6MV will be realized based on the acquisition of a CT-scan performed in treatment position. Intensity modulated RT (IMRT), volumetric modulated arc therapy (VMAT) and tomotherapy are authorized.
  W6: SURGERY Surgery should be performed as per Institutional practice by a surgeon with appropriate training in the treatment of sarcoma. The primary aim of surgery is to completely excise the tumor with a margin of normal tissue commonly accepted as 1 cm soft tissue, or equivalent
  W11 and W14: ATEZOLIZUMAB IV INJECTION. 2 injections of 1200 mg of atezolizumab with a 3-week interval
  Arms: pre-operative radiotherapy and post-operative atezolizumab

SUMMARY:
This multicentric, randomised, Phase II trial will use a pick-the-winner design in order to evaluate the clinical and biological activity of atezolizumab when combined with pre-operative or post-operative radiotherapy in STS patients.

Following Inform Consent Form (ICF) signature, eligible patients will be randomised (1:1:1) to receive:

* Arm A: Radiotherapy followed by atezolizumab then surgery.
* Arm B: Atezolizumab followed by surgery then radiotherapy.
* Arm C: Radiotherapy then surgery followed by atezolizumab.

The sequence of the study treatments is different among the 3 study arms. However, the dose regimens will be the same:

* Atezolizumab will be administered to all patients at the dose of 1200mg, by IV injection, for 2 cycles (Q3W).
* Radiotherapy will be administered to all patients at the dose of 2Gy/day, 5 days per week, for a total of 5 weeks and 50Gy.
* Surgery will be performed as per institutional practice.

Randomisation will be stratified according to histological subtypes as follows:

Group 1: Liposarcoma (LPS), Undifferentiated Pleomorphic Sarcoma (UPS), Leiomyosarcoma (LMS), myxofibrosarcoma, angiosarcoma versus Group 2: all translocation sarcoma except Ewing, rhabdomyosarcoma (RMS) and myxoid LPS.

DETAILED DESCRIPTION:
This trial is a European, multicenter, open-label, randomized, Phase II trial using a pick-the-winner design aiming to the clinical and biological activity of anti-PD-L1 (atezolizumab) in a population of operable localised soft tissue sarcomas (STS) patients to be treated with radiotherapy.

Following inform consent signature and validation of eligibility criteria, patients will be randomized (1:1:1) into one of the 3 study arms:

* Arm A: Pre-operative radiotherapy followed by 2 cycles of atezolizumab then surgery
* Arm B: 2 cycles of atezolizumab followed by surgery then post-operative radiotherapy
* Arm C: Pre-operative radiotherapy followed by surgery then 2 cycles of atezolizumab.

The sequence of treatment is different between the study arms, but the regimen of study treatments are the same. All randomized patients will received:

* The conventionally fractionated radiotherapy regimen of 2 Gy, 5 days a week up to a total dose of 50 Gy over 5 weeks. Radiotherapy will be either pre-(Arms A and C) or post-(Arm B) operative.
* Two cycles of atezolizumab (1200mg, IV, Q3W)
* Surgery will be performed as per institutional practice.

Randomisation will be stratified according to histological subtypes as follows

* Group 1: Leiomyosarcoma [LMS], Undifferentiated Pleomorphic Sarcoma [UPS], Liposarcoma [LPS], myxofibrosarcoma, angiosarcoma versus
* Group 2: all translocation sarcoma except Ewing, rhabdomyosarcoma RMS and myxoid LPS.

Following this sequence of treatment, all patients will be followed-up 2 weeks after the end of the treatment period then W18, W24 (=M6) then every 3 months until disease relapse, death, loss to follow-up. The minimal follow-up will be 1 year for the last randomized patient.

During the study period, the following tumor samples will be also collected for all randomized patients:

* A de novo tumor biopsy before study treatment start (pre-treatment tumor sample)
* A fragment of the surgery specimen.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 18 years at time of inform consent signature.
2. Histologically confirmed soft tissue sarcoma including liposarcoma, leiomyosarcoma, myxofibrosarcoma, UPS, angiosarcoma, all translocation sarcoma except Ewing, rhabdomyosarcoma (RMS), and myxoid liposarcoma (LPS).
3. Soft tissue sarcoma suitable for neoadjuvant RT and amenable to surgery with curative intent (high-grade non-metastatic tumors, intermediate and low-grade tumors greater than 5 cm).

   Note: Patients with local relapsing disease amenable to surgery are eligible.
4. Presence of at least one tumor lesion with a diameter ≥10 mm, visible by medical imaging and accessible to percutaneous or endoscopic sampling that permit core needle biopsy without unacceptable risk and suitable for retrieval of a minimum of three, but ideally 4, cores using a biopsy needle of at least 16-gauge.
5. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1 (Appendix 4).
6. Adequate end organs and bone marrow functions as defined below according to lab tests performed within 7 days before W1D1:

   * Bone marrow (without transfusion within 2 weeks before W1D1):

     * Hemoglobin ≥ 9.0 g/dL,
     * Absolute neutrophil count ≥ 1.5 x 109/L,
     * Platelets ≥ 100 x 109/L,
     * Lymphocyte count ≥ 0.5 x 109/L.
   * Renal function:

     * Serum creatinine clearance ≥ 30 mL/min/1.73m2 (MDRD or CKD-EPI formula - Appendix 3)
   * Hepatic function

     * Serum bilirubin < 1.5 × Upper Limit of Normal (ULN), with the following exception: Patients with known Gilbert disease who have serum bilirubin level ≤ 3 ULN may be enrolled.
     * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase ≤ 2.5 ULN.
   * Coagulation

     * INR and aPTT ≤ 1.5 ULN Note: This is applicable only for patients not receiving an anticoagulant treatment: patients receiving therapeutic anticoagulation must be on stable dose.
7. Minimal wash-out period for prior treatments (minimal time required from the end date of prior treatment to W1D1):

   * Immunosuppressive medication > 28 days, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid,
   * Live attenuated vaccines > 30 days, Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
   * Major surgical procedure, open biopsy (excluding skin cancer resection and screening tumor biopsy), or significant traumatic injury > 14 days (the wound must have healed),
   * Any approved or investigational anti-cancer therapy, including chemotherapy, hormonal therapy or targeted therapy > 21 days,
   * Systemic immunostimulatory agents > 28 days or five half-lives of the drug, whichever is longer,
   * Oral or IV antibiotics > 14 days.
8. Women of child-bearing potential must have a negative serum pregnancy test within 7 days before randomisation and must agree to use an effective form of contraception from the time of the negative pregnancy test up to 5 months after the last dose of atezolizumab (See Appendix 5).
9. Fertile men must agree to use an effective method of birth control during the study and for up to 5 months after the last dose of atezolizumab.
10. Patient should understand, sign, and date the written voluntary informed consent form prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.
11. Patients must be covered by a medical insurance in country where applicable.

Exclusion Criteria:

1. Patients with evidence of metastatic disease, defined by the presence of any of the followings:

   * Lesions that are discontinuous from the primary tumor,
   * Lesions that are not regional lymph nodes,
   * Lesions that do not share a body cavity with the primary tumor,
   * Evidence by medical imagining (eg CT-scan) of metastatic disease.
2. Patients with history of severe allergic or other hypersensitivity reactions to:

   * Chimeric or humanized antibodies or fusion proteins,
   * Biopharmaceuticals produced in Chinese hamster ovary cells, or
   * Any component of the atezolizumab formulation.
3. Patients using or requirement to use while on the study of any not permitted concomitant medications :

   * Any approved anti-cancer systemic treatment including chemotherapy, hormonotherapy, biological therapy, immunotherapy other than atezolizumab,
   * Any investigational agents,
   * Live vaccines. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, BCG, and typhoid (oral) vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however intranasal influenza vaccines (e.g. Flu-Mist®) are live attenuated vaccines, and are not allowed during the study active period,
   * Traditional herbal medicines since the ingredients of many herbal medicines are not fully studied and their use may result in unanticipated drug-drug interactions that may cause or confound assessment of toxicity,
   * Immunostimulatory agents, including but not limited to IFN-α, IFN-γ, or IL-2, during the entire study. These agents, in combination with atezolizumab, could potentially increase the risk for autoimmune conditions. In addition, all patients (including those who discontinue the study early) should not receive other immunostimulatory agents for 10 weeks after the last dose of atezolizumab,
   * Immunosuppressive medications, including but not limited to cyclophosphamide, azathioprine, methotrexate, and thalidomide. These agents could potentially alter the activity and the safety of atezolizumab. Systemic corticosteroids and anti-TNF-α agents may attenuate potential beneficial immunologic effects of treatment with atezolizumab but may be administered to manage irAE (See Safety Plan). If feasible, alternatives to these agents should be considered.
4. Patients with a malignancy other than STS within 5 years prior to randomisation with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome (such as adequately treated in situ carcinoma of the cervix, basal or squamous cell skin cancer, localised prostate cancer or ductal in situ carcinoma treated surgically with curative intent).
5. Patients with severe infections within 4 weeks prior to randomisation including but not limited to hospitalization for complications of infection, bacteraemia, or severe pneumonia.
6. Patients with history of autoimmune disease including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

   Note: Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:
   * Rash must cover less than 10% of body surface area (BSA).
   * Disease is well controlled at baseline and only requiring low potency topical steroids.
   * No acute exacerbations of underlying condition within the previous 12 months (not requiring PUVA [psoralen plus ultraviolet A radiation], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high-potency or oral steroids)" Note: Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible.

   Note: Patients with a type I diabetes well controlled by a stable dose of insulin are eligible.
7. Patients with active B or C hepatitis infection. Note: Patients with past Hepatitis B Virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. Patients positive for Hepatitis C Virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
8. Patients with active tuberculosis.
9. Patients with ongoing toxicities (Grade ≥1 according to CTCAE V5.0) from previous therapies, except for alopecia (any grades) and lab values defined in inclusion criteria.

   Note: Some Grade 2 may be permitted following discussion with the Sponsor.
10. Patients with evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including significant liver disease (such as cirrhosis, uncontrolled major seizure disorder, or superior vena cava syndrome).
11. Patients with significant cardiovascular disease, such as New York Heart Association cardiac disease Class II or greater, myocardial infarction within 3 months prior to W1D1, unstable arrhythmias or unstable angina.

    Notes:
    * Patients with a known Left Ventricular Ejection Fraction (LVEF) < 40% will be excluded
    * Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or LVEF < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
12. Patients with history of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e. bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on imaging.
13. Pregnant or lactating women.
14. Prior organ transplantation including allogeneic stem cell transplantation.
15. Patients who are known to be serologically positive for human immunodeficiency virus (HIV).

E16. Patient with prior treatment with anti-PD-1, or anti-PD-L1 immune checkpoint blockade therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathological impact of PD-L1 neutralisation (by atezolizumab) with or without radiotherapy versus radiotherapy alone in operable localised STS | 11 weeks
  Rate of pathological response (defined by at least 80°% of necrosis on surgery specimens) following PDL1 neutralisation with atezolizumab +/- radiotherapy versus RT alone

SECONDARY OUTCOMES:
Rate of patients with complete or near-complete pathologic response | 11 weeks
  Rate of patients with complete or near-complete pathologic response defined as ≥ 95% of necrosis. All pathology slides will be subjected to local central review by a subspecialty sarcoma pathologist. Surgery specimens will be examined for determination of tumor necrosis percentage.
Rate of patients with at least 50% of necrosis | 11 weeks
  Rate of patients with at least 50% of necrosis on the surgery specimen
Percentage of residual viable cells | 11 weeks
  Percentage of residual viable cells will be calculated for all surgery specimens.
Objective Response Rate (ORR) | 11 weeks
  Rate of patients with Complete Response (CR) and Partial Response (PR) as per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Tumor volume change | 11 weeks
  Tumor volume change (before versus after pre-operative treatment)
Quality of resection | 11 weeks
  Quality of resection will be described per study arms
Local Recurrence Rate (LRR) at 1 year post-surgery: | as long as 1 year from date of surgery
  Rate of local recurrence 1 year after surgery.
Time To Relapse (TTR) | from date of inclusion to relapse, for a maximum of 36 months from first randomized patient
  Time from inclusion to relapse of the disease.
Disease Free Survival (DFS) | Time after treatment ends that the patient survives without disease, for a maximum of 36 months from first randomized patient
  time alive without disease.
the impact of study treatments on immune cell infiltration | 11 weeks
  Number of T cells (including but not limited to GmzB+/CD8+ T-cell, CD3+ T-cell), B cells (CD20, IgG), and Treg (FOXP3) on pre (tumor biopsy at inclusion) and post-treatment (surgery specimen) by immunofluorescence (IF)
Number of patients with a significant change (at least a 2-fold change) in number of immune cell infiltration | 11 weeks
  Number of patients with a significant change (at least a 2-fold change) in number of T cells and other immune subsets under study treatments
Frequency of adverse events | a maximum of 36 months from date of first randomized patient
  Frequency of Adverse Event (AE), Serious Adverse Event (SAE), AE of special interest (AESI) and SUSAR graded using Common Terminology Criteria for Adverse Events (CTCAE) V4.03.
Amputation rate | 11 weeks
  Amputation rate will be measured per study arms
Severity of adverse events | a maximum of 36 months from date of first randomized patient
  Severity of Adverse Event (AE), Serious Adverse Event (SAE), AE of special interest (AESI) and SUSAR graded using Common Terminology Criteria for Adverse Events (CTCAE) V4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves BLAY, MD, Principal Investigator — Centre Leon Berard
Locations (6):
- France (5):
  - Institut Bergonie, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Royal Marsden Hospital, London, United Kingdom